CLINICAL TRIAL: NCT02008110
Title: A Randomized Controlled Trial of Carbohydrate Antigen 125-guided Therapy Among Patients Recently Discharged for Acute Heart Failure: Effect on 1-year Mortality or Readmission for Acute Heart Failure (CHANCE-HF).
Brief Title: Carbohydrate Antigen 125-guided Therapy in Heart Failure
Acronym: CHANCE-HF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundación para la Investigación del Hospital Clínico de Valencia (Other)
Collaborators: Ministerio de Sanidad, Servicios Sociales e Igualdad (Other Government)
Responsible Party: Principal Investigator, Julio Nuñez, MD, PhD, Fundación para la Investigación del Hospital Clínico de Valencia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EC10-108; 2011-000414-20 (EudraCT Number)
Record Dates: First submitted 2013-12-07; First posted 2013-12-11 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2016-02

CONDITIONS: Heart Failure
Keywords: Heart failure; Biomarker guided-therapy; Carbohydrate antigen 125; Clinical outcomes.
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CA125 guided strategy (Experimental): In this group, physician will be encouraged to maximize all treatment measures aimed to keep CA125≤35 U/ml (normal values).
  Interventions: Drug: CA125 guided strategy; Other: CA125 guided strategy
- Standard treatment strategy (Active Comparator): Therapy is based on established european current guidelines
  Interventions: Drug: Standard treatment strategy

INTERVENTIONS:
Drug: CA125 guided strategy — Up titration of loop diuretics according to plasma levels of CA125 in the active arm
  Arms: CA125 guided strategy
Drug: CA125 guided strategy — Consider statins in all patients in the active arm
  Arms: CA125 guided strategy
Drug: CA125 guided strategy — Consider omega-3 polyunsaturated fatty acids in the active arm
  Arms: CA125 guided strategy
Other: CA125 guided strategy — Frequency of monitoring according plasma evolution of CA125 in the active arm.
  Arms: CA125 guided strategy
Drug: Standard treatment strategy — All patients should be treated following standard european guidelines regarding angiotensin converting enzyme inhibitors, angiotensin receptor blockers, beta-blockers, aldosterone antagonists, diuretics, ivabradine and other treatments such as (diet, anticoagulants, antiarrhythmics, statins, omega-3 polyunsaturated fatty acids, digoxin, nitrates and vasoactive group).
  Arms: Standard treatment strategy
Drug: CA125 guided strategy — All patients should be treated following standard european guidelines regarding angiotensin converting enzyme inhibitors, angiotensin receptor blockers, beta-blockers, ivabradine and other treatments such as (diet, anticoagulants, antiarrhythmics, digoxin, nitrates and vasoactive group).
  Arms: CA125 guided strategy

SUMMARY:
Preliminary data suggest a potential role for monitoring and up-titrate pharmacological therapy of plasma levels of antigen carbohydrate 125 (CA125) following and admission for acute heart failure (AHF).

This study will evaluate the effect of a CA125-guided management strategy versus standard therapy on the composite endpoint of 1-year all-cause mortality or readmission for AHF in patients recently discharged for AHF.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older.
* At least 1 admission for AHF, in the last 180 days.
* Demonstrates functional New York Heart Association status of Class ≥II at the moment of enrollment.
* Objective evidence, either during the index admission or at least 180 days before enrollment, of a structural or functional abnormality of the heart at rest, and defined as: N terminal-pro-brain natriuretic peptide >1000 pg/ml or brain natriuretic peptide >100 pg/ml or echocardiographic abnormalities congruent with HF diagnosis such as: systolic left ventricular dysfunction (LVEF <50%); left ventricular hypertrophy (defined as left ventricular septum or left ventricular posterior wall thickness ≥12 millimeters or left ventricular mass index >104 g/m2 in women or 116 g/m2 in men); Ee'>15 or significant valvular heart disease (moderate-severe).
* A plasma CA125 value >35 U/ml in a recent test evaluation (at least 30 days before enrollment, and preferably assessed before hospital discharge).
* Patient must be capable of understanding and signing an informed consent form.

Exclusion Criteria:

* Life expectancy <12 months due to other diseases different from HF.
* Having undergone a cardiac transplantation, coronary revascularization procedure (percutaneous coronary intervention and/or coronary artery bypass grafting) or cardiac valve replacement in the past 3 months.
* Angina pectoris higher than class II (Canadian Cardiovascular Society Classification).
* Pregnancy at the moment of enrollment.
* Valvular heart disease already scheduled for surgical intervention.
* Severe chronic obstructive and/or restrictive pulmonary disease, requiring continuous oxygen administration.
* Serum creatinine level > 3 mg/dl or chronic renal insufficiency on dialysis treatment.
* Patients receiving resynchronization therapy during the index admission.
* Significant concurrent medical diseases including cancer or a history of cancer within 5 years of entering the screening period, endometriosis, cirrhosis, acute coronary syndrome within 6 months, uncontrolled hypertension, history of human immunodeficiency virus (HIV) infection, or a significant active infection.
* Participating in another randomized study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2011-12; Primary Completion 2014-07 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Composite of all-cause mortality plus acute heart failure related rehospitalization | 1 year

SECONDARY OUTCOMES:
Composite of total mortality plus readmission for any cause | 1 year
Days alive outside of the hospital | 1 year
Number of heart failure rehospitalizations. | 1 year
Number of episodes of worsening HF not requiring hospitalization | 1-year

CONTACTS AND LOCATIONS:
Overall Officials: Julio Núñez, MD, PhD, Principal Investigator — Fundación para la Investigación del Hospital Clínico de Valencia
Locations (1):
- Hospital Clínico Unbiversitario de Valencia, Valencia, Valencia, Spain

REFERENCES:
- [Derived] Nunez J, Llacer P, Bertomeu-Gonzalez V, Bosch MJ, Merlos P, Garcia-Blas S, Montagud V, Bodi V, Bertomeu-Martinez V, Pedrosa V, Mendizabal A, Cordero A, Gallego J, Palau P, Minana G, Santas E, Morell S, Llacer A, Chorro FJ, Sanchis J, Facila L; CHANCE-HF Investigators. Carbohydrate Antigen-125-Guided Therapy in Acute Heart Failure: CHANCE-HF: A Randomized Study. JACC Heart Fail. 2016 Nov;4(11):833-843. doi: 10.1016/j.jchf.2016.06.007. Epub 2016 Aug 10. PMID 27522630
- [Derived] Nunez J, Merlos P, Facila L, Llacer P, Bosch MJ, Bertomeu-Martinez V, Garcia-Blas S, Montagud V, Pedrosa V, Mendizabal A, Cordero A, Minana G, Sanchis J, Bertomeu-Gonzalez V; CHANCE-HF Investigators. Prognostic effect of carbohydrate antigen 125-guided therapy in patients recently discharged for acute heart failure (CHANCE-HF). Study design. Rev Esp Cardiol (Engl Ed). 2015 Feb;68(2):121-8. doi: 10.1016/j.rec.2014.03.018. Epub 2014 Aug 10. PMID 25623430